CLINICAL TRIAL: NCT01378013
Title: Metabolic Phenotyping and Systems Biology in Surgery
Brief Title: SurgicAl Metabolic Phenotyping Longitudinal Evaluation Study
Acronym: SaMPLE
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 11/L0/686; NIHR BRC (Other Grant/Funding Number: P31675)
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2011-07

CONDITIONS: Colon Cancer; Breast Cancer; Trauma; Inflammatory Bowel Disease; Hernia
Keywords: Metabonomics; Systems biology; Intelligent knife; Colorectal cancer; NMR; Mass spectrometry
MeSH Terms: conditions — Colonic Neoplasms; Breast Neoplasms; Wounds and Injuries; Inflammatory Bowel Diseases; Hernia; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Urine
  2. Blood (plasma)
  3. Stool / small bowel content
  4. Tissue (Colon, small bowel,stomach,eosophagus, breast, lymph nodes)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Elective sugery: Patients entering into elective surgery. These will be divided into three subgroups:
  A. Patients with cancer. This will include patients with malignancy of the gastrointestinal and colorectal tract (including those excised by microsurgery) cancer of the breast or solid tumours of the kidney.
  B. Patients with benign diseases of the bowel requiring surgery e.g. inflammatory bowel disease C. Benign surgical conditions, usually operated on in a day surgery setting. These will specifically be of the biliary tree (gall stones) and the anterior abdominal wall (e.g. Hernia surgery)
- Acute (emergency) surgery: Patients presenting to Accident and emergency under the care of the general surgery on call team will be recruited into this study group. This study group will have the following subgroups:
  A. Acute abdominal pain, as per the previous ethical clearance B. Patients with acute sepsis thought to be of surgical origin. C. Patients suffering major trauma with an Injury severity score of >15, multiple injuries, who require surgery or who have >1 organ system that is failed or who are admitted to the intensive care department.

SUMMARY:
This work will use a new approach to measure how surgery effects human biochemistry and metabolism. It will create a metabolic signature or 'phenotype' for surgical injury that will help clinicians choose the right surgical treatments for an individual. This is because metabolism is based on an individual's genes, disease burden and environmental influences such as gut microbiota. This study will use a scientific method based on computational analysis of spectra taken from techniques known as Mass Spectrometry (MS) and Nuclear Magnetic Resonance (NMR) spectroscopy. This science is called 'metabonomics' and it has many advantages. Firstly, it provides a measure of thousands of metabolites at a single moment in time that are unique to the individual and it therefore gives a 'systems' overview of a persons metabolism. Secondly it is able to process many hundreds of samples quickly. The investigators are aiming to integrate the investigators metabolic data with genetic information about patients or bacteria wherever possible. This will be the first time that a 'systems biology' approach has been used in surgery, with potentially significant gains to me made in pre operative risk stratification and optimisation. By performing this analysis at all stages of the surgical journey (preoperatively, during the operation and after the surgery) it will ensure the right treatments are given to the right patient at the right time. By creating longitudinal models of the biochemical responses to surgery, predict at a much earlier stage those patients at risk of developing complications. This will improve outcome after surgery. This work will use a metabonomic approach to create new tools for surgeons to use during operations based on tissue biology. For example the investigators will be able to measure the metabolic content of tumours in real time by measuring the biological content of diathermy smoke. This has the potential to change intra-operative decision making and further improve outcome.

DETAILED DESCRIPTION:
A systems perspective can improve surgical decision making both before and after surgery in real time. Specifically, we hypothesize that it may provide diagnostic and prognostic information of importance that is more accurate than current biochemical approaches. This is because it accounts for important environmental influences on surgical outcome such as pharmacotherapy and the gut microbiota.

The secondary hypothesis is that this approach can provide real time molecular feedback to the operator during surgery about tissue type and pathology.

This work will therefore need to study patients having surgery under a range of different conditions and states, and by varying types of surgical intervention. It is known that patients with cancer for example have quite different metabolic requirements to those without. This has significant implications for the development of personalized management strategies for patients with cancer undergoing surgery. It is essential that this study definitively proves that the technology is able to make a description between patients with significantly different disease states and also that it can differentiate this from the type and magnitude of the surgical procedure being performed and the timing of the surgery. Therefore, this work will involve a heterogeneous patient cohort.

Study design:

This study will be subject to research governance structures provided internally within the department of Biosurgery and Surgical technology in conjunction with the section of Biomolecular medicine for the safe use of samples and machinery. It will also possess a clinical steering committee to assess the progress, clinical outcomes, safety and timely completion of the work.

Two separate clinical groups will be recruited for this trial. The first will be those patients undergoing elective procedures, the second will be those undergoing emergency procedures. Each of these groups will contain subcategories of clinical conditions, upon which the study will focus.

Elective surgery (n=200):

A. Patients with cancer. This will include patients with malignancy of the gastrointestinal and colorectal tract (including those excised by microsurgery) cancer of the breast or solid tumors of the kidney.

B. Patients with benign diseases of the bowel requiring surgery e.g. inflammatory bowel disease C. Benign surgical conditions, usually operated on in a day surgery setting. These will specifically be of the biliary tree (gall stones) and the anterior abdominal wall (e.g. Hernia surgery)

Patients will be recruited if seen under the 'two week' wait rule with suspected cancer for the general surgery, upper GI surgery, Breast and Urology surgery teams at St. Mary's hospital in the outpatient setting.

Patients attending for elective inpatient surgery under the general, upper GI or breast surgery teams at St. Mary's hospital, London will be recruited at the pre admission clinic.

Acute surgery (n=200)

Patients presenting to Accident and emergency under the care of the general surgery on call team will be recruited into this study group. This study group will have the following subgroups:

A. Acute abdominal pain, as per the previous ethical clearance B. Patients with acute sepsis thought to be of surgical origin. C. Patients suffering major trauma with an Injury severity score of >15, multiple injuries, who require surgery or who have >1 organ system that is failed or who are admitted to the intensive care department.

Exclusion criteria:

All patients under the age of 18 years All patients who are pregnant Patients receiving Advanced Life Support by cardiopulmonary resuscitation on their arrival in hospital.

Patients with advanced cancer only suitable for palliative care at presentation to the clinical team.

Patients presenting for the first time with other known malignancies for which they are receiving treatment e.g. Prostate cancer Patients already recruited into other clinical studies.

This study will be broken down into two separate phases:

Preclinical work:

Preclinical work for biofluid analysis in elective and acute surgical admissions has already been performed in both animal and human studies in Magic Angle Spinning (MAS)-1H NMR (also known as solid state NMR as the tissue does not require preparation), MS, and Matrix Assisted Laser Desorption Ionization (MALDI)-MS. Samples from previous studies gained under ethical clearance will be analyzed using these techniques for methodological optimization. This will entail metabonomic and metagenomic profiling of colorectal cancer samples (Ethics Ref: 07/H0712/112 and 06/Q0403/16) and from samples taken from patients with acute pancreatitis and the acute abdomen (Ethics Ref: 05/Q0403/201).

Non essential (i.e. Benign or pathologically normal tissue) excised and due for incineration taken from consenting patients during routine surgery will be collected for analysis by: Mass spectrometry of smoke plumes collected from a range of electrocautery devices. This will allow optimization of MS protocols and it will define the chemical parameters for normal tissue and for various tissue types.

b. Malignant tissue excised from breast, colon and upper GI cancers will be tested for its capacity to detect normal and malignant disease by the use of the intelligent knife ex vivo. This will be performed under the guidance of histopathologists, and it will not interfere with pathological staging or treatment of cancers.

Development of translational software for analytical interpretation of complex biochemical metadata by non scientific staff will be developed using these data. This work will use current intensive care clinical databases.

Clinical work:

The aim is for the technology to be readily applicable to patients having surgery within the NHS. Therefore, patients will be recruited from two surgical pathways:

Acute Care: Patient recruitment

Patients will be recruited whilst in Accident and Emergency. Only patients admitted via this route will be eligible for study inclusion. Patients will be provided with an information sheet and the patient will be left for 30 minutes to consider the study. Consent will be taken in private, by an adequately qualified and trained individual. When consented, patients will be asked to complete a questionnaire to provide medical and surgical history, and metabolic information that could influence results.

It will not be possible to gain consent in some cases as patients may be unconscious or unable to consent due to injury. In these cases samples will be taken, and when the patient gains consciousness and capacity formal consent will be taken. If at this stage, the patient states they do not want to be included in the study their samples will be withdrawn. In the event of a patient's death, the samples will be included in the study. This is because the capacity of these tests to predict mortality is a primary end point.

Elective Care: Patient recruitment

Patients will be recruited in the outpatient setting where ever possible to ensure that they have adequate time to take on board the clinical information and to consent. We will sample patients on their admission to hospital for treatment after the decision for surgery has been made.

Sample Collection:

Samples will be collected at set time points during the patient journey in both cases. Samples will be obtained at the same time as standard clinical investigations to minimize discomfort for the patient, and they will not be taken in excess of standard sample times prevent unnecessary investigation for the patient. Sample collection will be coordinated with the clinical biochemistry team at St. Mary's hospital where ever possible to prevent unnecessary and time consuming sampling.

Pre operation:

Plasma and urine collection:

1. At their arrival in Accident and Emergency. Every 24 hours for the duration of their admission or until surgery, discharge or treatment defined as surgical, radiological or invasive therapeutic intervention.

If the patient remains in hospital for prolonged rehabilitation or non surgical therapy, samples will be taken weekly until discharge.

Stool sample

First bowel motion after arrival in A+E. Preoperative and pre bowel preparation sample before surgery. This will be given either in clinic or on the ward.

Tissue sample collection

Preoperative biopsy

In the event that patients are sent for routine endoscopic or biopsy, samples of tissue will be taken for metabonomic analysis.

b. Intra-operative.

Analysis of smoke plumes by MS will be performed for each case. This will not interfere with the standard operation and the operating surgeon will not be asked to make a decision based on the data from the experiment. In cases of cancer resections, tissue samples will be collected in keeping within the principals of oncological surgery. In the cases of breast surgery, sentinel lymph nodes will also be harvested and analyzed by NMR. During colorectal surgery, tissue from the mesorectum will be taken for analysis from standard collection points and in upper GI cancer resections, similar principals will apply for sampling. In acute or emergency situations, tissue will also be taken from areas of tissue thought to be at risk of ischemia (e.g. anastomotic sites were bowel is to be joined).

Stool and small bowel effluent will be harvested at the time of surgery so that the effect of surgery on the gut microbial ecosystem can also be accounted for.

c. Post operative.

Urine and plasma will be sampled daily post operatively in keeping with current clinical practice for the first week. Where ever possible, no extra samples will be collected beyond those sampled by the clinical staff.

Stool samples will also be collected. The first bowel motion will be collected after surgery, and then each motion until the first week is completed, and then weekly after this.

The first motion from stoma / ileostomy: If stoma sited, daily samples will be taken for the first week.

Weekly samples will then be collected until discharge.

In the event that a patient returns to theatre, the sample collection sequence will re commence.

All clinical data will be recorded for the duration of the patient stay. This will refer to pre operative information and assessment where possible, physiological data, radiological findings, clinical biochemistry, surgical and clinical outcome and length of stay. This will be anonymous and coded.

On discharge, patients will be bought back to clinic at 8 weeks for clinical assessment as per the routine analysis. Samples of urine, blood and stool will be taken at this time. Oncological patients will be followed up for five years as per the oncology protocol at St. Mary's Hospital Paddington.

ELIGIBILITY:
Inclusion Criteria:

1. Elective surgery (n=200)

   * Patients with cancer. This will include patients with malignancy of the gastrointestinal and colorectal tract (including those excised by microsurgery)cancer of the breast or solid tumours of the kidney.
   * Patients with benign disease of the bowel requiring surgery e.g. inflammatory bowel disease
   * Benign surgical conditions, usually operated on in a day surgery setting. These will specifically be of the biliary tree (gall stones) and the anterior abdominal wall (e.g. Hernia surgery)
   * Patients will be recruited if seen under the 'two week' wait rule with suspected cancer for the general surgery, upper GI surgery, Breast and Urology surgery teams at St. Mary's hospital in the outpatient setting will be recruited
   * Patients attending for elective inpatient surgery under the general, upper GI or breast surgery teams at St. Mary's hospital, London will be recruited at the pre admission clinic.
2. Acute surgery (n=200) Patients presenting to Accident and emergency under the care of the general surgery on call team will be recruited into this study group. This study group will have the following subgroups:

   * Acute abdominal pain
   * Patients with acute sepsis thought to be of surgical origin as diagnosed by their history, clinical examination and routine investigations.
   * Patients suffering major trauma with an Injury severity score (ISS) of >15, multiple injuries, who require surgery or who have >1 organ system that is failed or who are admitted to the intensive care department.

Exclusion Criteria:

* All patients under the age of 18 years
* All patients who are pregnant
* Patients receiving Advanced Life Support by cardiopulmonary resuscitation on their arrival in hospital.
* Patients with advanced cancer only suitable for palliative care at presentation to the clinical team.
* Patients presenting for the first time with other known malignancies for which they are receiving treatment e.g. Prostate cancer
* Patients already recruited into other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two separate clinical groups will be recruited for this trial. The first will be those patients undergoing elective procedures, the second will be those undergoing emergency procedures.
  Elective surgery (n=200):
  Acute surgery (n=200)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-08; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Sepsis | 30 days
  Daily sampling of patients during the post operative period to determine early biomarkers for the development of sepsis

SECONDARY OUTCOMES:
Oncological resection margins | 10 days
  All resected cancers will be done so using the intelligent knife. Samples will be analysed by histology as per standard clinical practice. It will be determined if the intelligent knife can reduce positive resection margins.
Local and distant recurrence | 5 years
  To determine if long term metabonomic phenotyping can predict both local and distant recurrence after oncological recurrence of cancers.
Organ failure | 30 days
  We will determine novel biomarkers for predicting organ failure after injury (trauma) and surgery
Mortality | 30 days
  This study will determine whether a systems biology approach can predict mortality before other routinely used clinical biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Ara W Darzi, PC, KBE, Principal Investigator — Imperial College London; Jeremy K Nicholson, FMedSci, Study Director — Imperial College London; Elaine Holmes, PhD, Study Chair — Imperial College London
Locations (1):
- Department of BioSurgery and Surgical Technology, Imperial College London, London, London, United Kingdom

REFERENCES:
- [Background] Kinross JM, Holmes E, Darzi AW, Nicholson JK. Metabolic phenotyping for monitoring surgical patients. Lancet. 2011 May 28;377(9780):1817-9. doi: 10.1016/S0140-6736(11)60171-2. Epub 2011 May 17. No abstract available. PMID 21596428
- [Background] Li JV, Ashrafian H, Bueter M, Kinross J, Sands C, le Roux CW, Bloom SR, Darzi A, Athanasiou T, Marchesi JR, Nicholson JK, Holmes E. Metabolic surgery profoundly influences gut microbial-host metabolic cross-talk. Gut. 2011 Sep;60(9):1214-23. doi: 10.1136/gut.2010.234708. Epub 2011 May 14. PMID 21572120
- [Background] Kinross JM, Darzi AW, Nicholson JK. Gut microbiome-host interactions in health and disease. Genome Med. 2011 Mar 4;3(3):14. doi: 10.1186/gm228. PMID 21392406
- [Background] Kinross JM, Alkhamesi N, Barton RH, Silk DB, Yap IK, Darzi AW, Holmes E, Nicholson JK. Global metabolic phenotyping in an experimental laparotomy model of surgical trauma. J Proteome Res. 2011 Jan 7;10(1):277-87. doi: 10.1021/pr1003278. Epub 2010 Nov 24. PMID 21105667
- [Background] Kinross J, von Roon AC, Penney N, Holmes E, Silk D, Nicholson JK, Darzi A. The gut microbiota as a target for improved surgical outcome and improved patient care. Curr Pharm Des. 2009;15(13):1537-45. doi: 10.2174/138161209788168119. PMID 19442171
- [Background] Nicholson JK, Wilson ID, Lindon JC. Pharmacometabonomics as an effector for personalized medicine. Pharmacogenomics. 2011 Jan;12(1):103-11. doi: 10.2217/pgs.10.157. PMID 21174625
- [Background] Beckonert O, Coen M, Keun HC, Wang Y, Ebbels TM, Holmes E, Lindon JC, Nicholson JK. High-resolution magic-angle-spinning NMR spectroscopy for metabolic profiling of intact tissues. Nat Protoc. 2010 Jun;5(6):1019-32. doi: 10.1038/nprot.2010.45. Epub 2010 May 13. PMID 20539278
- [Background] Lucas C, Jenkins P, Mendels J, Due D, Forbes WP, Sirgo MA. The effectiveness of labetalol compared to hydrochlorothiazide in hypertensive black patients. J Natl Med Assoc. 1991 Oct;83(10):866-71. PMID 1800760
- [Background] Duarte IF, Stanley EG, Holmes E, Lindon JC, Gil AM, Tang H, Ferdinand R, McKee CG, Nicholson JK, Vilca-Melendez H, Heaton N, Murphy GM. Metabolic assessment of human liver transplants from biopsy samples at the donor and recipient stages using high-resolution magic angle spinning 1H NMR spectroscopy. Anal Chem. 2005 Sep 1;77(17):5570-8. doi: 10.1021/ac050455c. PMID 16131067
- See also: Division of surgery, Imperial College London — http://www1.imperial.ac.uk/surgeryandcancer/divisionofsurgery/biomol_med/